CLINICAL TRIAL: NCT03218618
Title: CHOKing Prevention Project
Acronym: CHOP
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Other Study IDs: CHOP2017
Record Dates: First submitted 2017-06-01; First posted 2017-07-14 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Health Knowledge; Attitudes; Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of such study is to compare three different school-based (in nurseries, kindergartens and primary schools) interventions aimed at teaching to families how to prevent food choking injuries.

The topic of food choking primary and secondary prevention is placed in a more general topic regarding food safety, including education on food labeling and on food waste prevention.

DETAILED DESCRIPTION:
The CHOP has been designed as a community intervention trial that compares three different school-based intervention strategies aimed at teaching to families how to prevent food choking injuries in children, together with the basics of food safety. The choice of employing such study design is motivated by the facts that community intervention trials allow to reach as many people as possible regardless their risk of experiencing the outcome of interest and to inform policy-makers on the effectiveness of an intervention on a community basis instead of an individual basis.

Forty-eight educational facilities (nurseries, kindergartens and primary schools) equally distributed between North, Centre, South, and major Islands of Italy will be enrolled.

Educational facilities will be stratified so that each stratum will include one educational facility from each educational stage (stratum=1 nursery, 1 kindergarten, 1 primary school).

The assessment of the effectiveness of each intervention strategy will be performed through a structured telephonic interview one month after the delivery of the intervention. I

Schools, to be enrolled, must provide:

* availability of at least 45 families (one member from each family will be involved in the study);
* availability of a room and of technological system (monitor, sound system) allowing the performance of the educational intervention;
* availability of administrative support;
* approval of the inclusion in the study by school's competent bodies.

Family members (one from each family) must be:

* aged >18 years;
* parent of children attending the school or person exercising the parental authority on children attending the school;
* without physical impairments not allowing the performance of practical activities;
* willing to participate at all stages of the study;
* signed informed consent.

ELIGIBILITY:
Inclusion Criteria:

-

Schools, to be enrolled, must provide:

* availability of at least 45 families (one member from each family will be involved in the study);
* availability of a room and of technological system (monitor, sound system) allowing the performance of the educational intervention;
* availability of administrative support;
* approval of the inclusion in the study by school's competent bodies.

Family members (one from each family) must be:

* aged >18 years;
* parent of children attending the school or person exercising the parental authority on children attending the school;
* without physical impairments not allowing the performance of practical activities;
* willing to participate at all stages of the study;
* signed informed consent.

Exclusion Criteria:

* Schools that will not meet inclusion criteria will not be enrolled in the study.

Family members who will not meet the inclusion criteria will not be involved in the study.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Families
Sampling Method: Probability Sample
Enrollment: 1670 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
percentage of correct answers to telephonic structured interview | up to 30 days after the intervention
  percentage (%)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Padova, Padua, PD, Italy

REFERENCES:
- [Derived] Lorenzoni G, Azzolina D, Baldas S, Messi G, Lanera C, French MA, Da Dalt L, Gregori D. Increasing awareness of food-choking and nutrition in children through education of caregivers: the CHOP community intervention trial study protocol. BMC Public Health. 2019 Aug 22;19(1):1156. doi: 10.1186/s12889-019-7469-7. PMID 31438901